CLINICAL TRIAL: NCT02998476
Title: A Phase 2, Multicenter, International, Open-Label, Safety and Efficacy Study of INCB050465 in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (CITADEL-202)
Brief Title: A Phase 2 Safety and Efficacy Study of INCB050465 in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (CITADEL-202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-202/CITADEL-202; Parsaclisib (Other: Incyte Corporation); 2016-002205-19 (EudraCT Number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: Diffuse large B-cell lymphoma; relapsed; refractory; non-Hodgkin lymphoma; phosphatidylinositol 3-kinase δ (PI3Kδ) inhibitor; Bruton's tyrosine kinase (BTK)
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Non-Hodgkin | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A Parsaclisib (no prior BTK inhibitor) (Experimental): Parsaclisib in subjects who were not previously treated with a BTK inhibitor.
  Interventions: Drug: Parsaclisib
- Group B Parsaclisib (prior BTK inhibitor) (Experimental): Parsaclisib in subjects who were previously treated with a BTK inhibitor.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib once daily for 8 weeks followed by once weekly
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to assess the safety and efficacy of parsaclisib in subjects with relapsed or refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Eligible 19 years and older in South Korea
* Relapsed or refractory DLBCL, which has been histologically documented, defined as having received at least 2 but no more than 5 prior treatment regimens and ineligible for high-dose chemotherapy supported by autologous stem cell transplant.
* Must have ≥ 1 measurable lesion (≥2 cm in longest dimension) or ≥ 1 measurable extranodal lesion (≥1 cm in longest dimension) on computed tomography (CT) scan or magnetic resonance imaging (MRI).
* Subjects must be willing to undergo an incisional or excisional lymph node biopsy of accessible adenopathy or provide the most recent, available archived tumor biopsy.
* Eastern Cooperative Oncology Group performance status 0 to 2.

Exclusion Criteria:

* Primary mediastinal (thymic) large B-cell lymphoma.
* Known brain or central nervous system metastases or history of uncontrolled seizures.
* Allogeneic stem cell transplant within the last 6 months, or active graft versus host disease following allogeneic transplant, or autologous stem cell transplant within the last 3 months.
* Use or expected use during the study of any prohibited medications, including potent cytochrome P450 3A4 inhibitors or inducers within 14 days or 5 half lives (whichever is longer) before the first dose of study drug.
* Prior treatment with the following:

  * Group A: Prior treatment with a selective phosphatidylinositol 3-kinase (PI3K) δ inhibitor (eg, idelalisib), a pan-PI3K inhibitor, or a BTK inhibitor (eg, ibrutinib).
  * Group B: Prior treatment with a selective PI3Kδ inhibitor (eg, idelalisib) or a pan PI3K inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Corrado, MD, Study Director — Incyte Corporation
Locations (70):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Sutter Gould Medical Foundation, Modesto, California
  - Sharp Memorial Hospital, San Diego, California
  - Advanced Pharma CR, LLC, Miami, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Advocate Medical Group Niles Milwaukee Ave, Niles, Illinois
  - Indiana BMT, Beech Grove, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Kentucky Hospital, Lexington, Kentucky
  - St. Agnes Hospital, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - CHI Health - St. Francis Medical Center, Grand Island, Nebraska
  - Summit Medical Group, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Utah Cancer Specialists- Network, Salt Lake City, Utah
- Australia (6):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (4):
  - ZNA Stuivenberg, Antwerp
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- LHSC - Victoria Hospital, London, Ontario, Canada
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - Fakultni nemocnice v Motole, Prague
- France (14):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Centre Francois Baclesse, Caen, Calvados
  - CHU Dijon - Hopital du Bocage, Dijon, Cote dÝOr
  - Centre Hospitalier Libourne, Libourne, Gironde
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble, Isere
  - Centre Hospitalier d'Angers, Angers, Maine Et Loire
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hôpital Saint-Louis, Paris, Paris
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Chu de Grenoble - Hopital Albert Michallon, Grenoble
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Chu Vandoeuvre-Les-Nancy Hopital Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
- Poland (3):
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Malopolskie Centrum Medyczne s.c., Krakow
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - ICO l´Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Txagorritxu, Vitoria-Gasteiz
- United Kingdom (3):
  - The Christie, Manchester, Greater Manchester
  - Southend University Hospital, Southend-on-Sea
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Coleman M, Belada D, Casasnovas RO, Gressin R, Lee HP, Mehta A, Munoz J, Verhoef G, Corrado C, DeMarini DJ, Zhao W, Li J, Fay K. Phase 2 study of parsaclisib (INCB050465), a highly selective, next-generation PI3Kdelta inhibitor, in relapsed or refractory diffuse large B-cell lymphoma (CITADEL-202). Leuk Lymphoma. 2021 Feb;62(2):368-376. doi: 10.1080/10428194.2020.1832660. Epub 2020 Nov 3. PMID 33140664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase 2, multicenter, international, open-label study with approximately 120 planned participants with relapsed or refractory DLBCL.
Pre-assignment Details: 55 participants included in the treatment group A who were not previously treated with a BTK inhibitor and received parsaclisib 20 mg QD for 8 weeks followed by 20 mg QW. 5 Participants were enrolled in group B who were previously treated with a BTK inhibitor. and received parsaclisib 20 mg QD for 8 weeks followed by 20 mg QW.
Period: Overall Study
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor) | Group B Parsaclisib (Prior BTK Inhibitor)
Started (60) | 55 | 5
Completed (0) | 0 | 0
Not Completed | 55 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participants transferred to rollover study INCB50465-801 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 45 | 2
Not completed — Other | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor) | Group B Parsaclisib (Prior BTK Inhibitor) | Total
Number analyzed (Participants) | 55 | 5 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (12.62) | 68.4 (12.97) | 69.5 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 0 | 22
  Male | 33 | 5 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 42 | 5 | 47
  Black or African American | 2 | 0 | 2
  Asian | 3 | 0 | 3
  Other | 6 | 0 | 6
  Missing | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 37 | 5 | 42
  Not Reported | 10 | 0 | 10
  Unknown | 7 | 0 | 7
  Missing | 1 | 0 | 1
ECOG [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) scale describes a patient's level of functioning in terms of their ability to care for themselves, activity, and ability. The scale is from 0 to 5; 0 - Fully active; 1 - Restricted in physically strenuous activity but ambulatory; 2- Ambulatory and capable of all selfcare but unable to carry out any work activities; 3- Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; 5 - Dead.
  Participants
    0 | 12 | 1 | 13
    1 | 34 | 3 | 37
    2 | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Based on Lugano Classification Criteria in Group A
Description: Defined as the percentage of subjects with a complete or partial response as defined by Lugano Classification criteria for lymphomas (Cheson et al 2014) as determined by IRC.
Time Frame: Every 9 weeks through Week 27, then every 18 weeks thereafter until disease progression, up to 26 months
Population: The full analysis set includes all subjects enrolled in the study who received at least 1 dose of INCB050465
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor)
Number analyzed (Participants) | 55
percentage | 25.5 [14.7 to 39.0]

2. Secondary Outcome: Duration of Response in Group A
Description: Defined as the time from first documented evidence of complete or partial response until disease progression or death from any cause among subjects who achieve an objective response as determined by IRC.
Time Frame: Every 9 weeks through Week 27, then every 18 weeks thereafter until disease progression, up to 26 months
Population: The full analysis set includes all subjects enrolled in the study who received at least 1 dose of INCB050465
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor)
Number analyzed (Participants) | 55
months | 6.2 [2.1 to NA] — The upper boundary of the 95% CI was not reached

3. Secondary Outcome: Progression-free Survival in Group A
Description: Defined as the time from the date of the first dose of study drug until the earliest date of disease progression, as determined by radiographic disease assessment as provided by an IRC.
Time Frame: Every 9 weeks through Week 27, then every 18 weeks thereafter until disease progression, up to 26 months
Population: The full analysis set includes all subjects enrolled in the study who received at least 1 dose of INCB050465
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor)
Number analyzed (Participants) | 55
months | 2.2 [2.0 to 4.1]

4. Secondary Outcome: Overall Survival (OS) in Group A
Description: Defined as the time from the date of the first dose of study drug until death by any cause.
Time Frame: From first dose of study drug until death by any cause; up to 26 months
Population: The full analysis set includes all subjects enrolled in the study who received at least 1 dose of INCB050465
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor)
Number analyzed (Participants) | 55
months | 7.0 [3.5 to NA] — The upper boundary of the 95% CI was not reached

5. Secondary Outcome: Safety as Assessed by Percentage of Subjects With Adverse Events in Group A and Group B
Description: A TEAE is any AE either reported for the first time or worsening of a pre-existing event after the first dose of parsaclisib until 30 days after the last dose administration.
Time Frame: Screening through 35 days after end of treatment, up to 42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor) | Group B Parsaclisib (Prior BTK Inhibitor)
Number analyzed (Participants) | 55 | 5
Participants | 50 | 4

ADVERSE EVENTS:
Time Frame: Screening through 35 days after end of treatment, up to 42 months
Groups:
- Total: Total
Arm/Group | Group A Parsaclisib (no Prior BTK Inhibitor) | Group B Parsaclisib (Prior BTK Inhibitor) | Total
All-Cause Mortality (participants affected / at risk) | 45/55 | 3/5 | 48/60
Serious Adverse Events (participants affected / at risk) | 39/55 | 2/5 | 41/60
Other Adverse Events (participants affected / at risk) | 41/55 | 3/5 | 44/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Parsaclisib (no Prior BTK Inhibitor) (N=55) | Group B Parsaclisib (Prior BTK Inhibitor) (N=5) | Total (N=60)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (3) | 0 (0) | 1 (3)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (8) | 0 (0) | 5 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Parsaclisib (no Prior BTK Inhibitor) (N=55) | Group B Parsaclisib (Prior BTK Inhibitor) (N=5) | Total (N=60)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 0 (0) | 4 (6)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0) | 9 (10)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 0 (0) | 10 (11)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (2) | 8 (9)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 4 (4)
Fatigue (General disorders) | 4 (4) | 1 (1) | 5 (5)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (3) | 1 (1) | 2 (4)
Nausea (Gastrointestinal disorders) | 11 (11) | 0 (0) | 11 (11)
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 4 (5)
Pyrexia (General disorders) | 5 (7) | 0 (0) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0) | 4 (5)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02998476/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02998476/SAP_001.pdf